CLINICAL TRIAL: NCT01929018
Title: Collaborative-care Rehabilitation to Improve Functional Outcomes After Dysvascular Amputation
Brief Title: Collaborative-care Rehabilitation After Dysvascular Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0179
Record Dates: First submitted 2013-08-19; First posted 2013-08-27 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Complications; Peripheral Arterial Disease
Keywords: Amputation; Rehabilitation; Exercise; Movement
MeSH Terms: conditions — Diabetes Complications; Peripheral Arterial Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise, activity, and self-management (Experimental): Exercise, Walking Program, and Health Self-Management Support. Participants will be visited at home once monthly and contacted by phone once weekly over 12 weeks to deliver the interventions.
  Interventions: Behavioral: Exercise; Behavioral: Walking Program; Behavioral: Health Self-Management Support
- Home and phone visit (No Intervention): No intervention will be applied. Participants will be visited at home once monthly and contacted by phone once weekly over 12 weeks to monitor health status.

INTERVENTIONS:
Behavioral: Exercise — Exercise will target muscle strength and joint mobility impairments and will be delivered over a 12 week period.
  Arms: Exercise, activity, and self-management
Behavioral: Walking Program — A walking program will be established with the goal of participants walking at least five days per week. Duration of program is 12 weeks.
  Arms: Exercise, activity, and self-management
Behavioral: Health Self-Management Support — Health self-management support will be delivered with weekly meetings between the researcher and participant over a 12-week period.
  Arms: Exercise, activity, and self-management

SUMMARY:
The objective of this study is to examine the feasibility of using a collaborative-care, home-based rehabilitation program to improve functional outcomes for people recovering from lower limb amputation caused by vascular problems and/or diabetes complications. The primary hypothesis is that the rehabilitation program will result in greater improvements in performance-based and participant-reported measures of physical function, compared to standard of care after outpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes and/or Peripheral Artery Disease
2. Unilateral transtibial amputation < 6 months prior to screening
3. Household ambulation using definitive prosthesis prior to baseline testing
4. Participation in physical rehabilitation at time of baseline testing
5. Live within 45 minutes of a participating clinic

Exclusion Criteria:

1. Require wheelchair for mobility (use prosthesis for transfers only)
2. Ankle-level or above amputation on contralateral limb
3. Traumatic or cancer-related amputation
4. Uncontrolled heart condition
5. Acute systemic infection
6. Pregnancy
7. Decisionally challenged
8. Prisoners

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory L Christiansen, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Christiansen CL, Miller MJ, Murray AM, Stephenson RO, Stevens-Lapsley JE, Hiatt WR, Schenkman ML. Behavior-Change Intervention Targeting Physical Function, Walking, and Disability After Dysvascular Amputation: A Randomized Controlled Pilot Trial. Arch Phys Med Rehabil. 2018 Nov;99(11):2160-2167. doi: 10.1016/j.apmr.2018.04.011. Epub 2018 May 7. PMID 29746823

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant study events occurred after participants were enrolled, but before they were assigned to a study group.
Period: Overall Study
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Hospitalization | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (6.0) | 65 (11.3) | 63.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 16 | 19 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 38
Site of Rehab, n, Veterans Administration Medical Center [Count of Participants; unit: Participants] — Number of participants treated at Veterans Administration Medical Center
  Participants | 10 | 10 | 20
BMI, kg/m2 [Mean (Standard Deviation); unit: kg/m^2] | 31 (10.6) | 30 (6.3) | 31 (8.6)
Time Since Amputation, weeks [Mean (Standard Deviation); unit: weeks] | 16 (6.5) | 20 (6.4) | 18 (6.6)
Geriatric Depression Scale, score out of 15 [Mean (Standard Deviation); unit: units on a scale] — Scale range is 0-15. Score is total out of possible maximum of 15. A score of 0 to 5 is normal. A score greater than 5 suggests referral for assessment of depression.
  units on a scale | 2.8 (3.2) | 3.2 (2.6) | 3.0 (2.9)
Mini Mental Status Exam, score out of 30 [Mean (Standard Deviation); unit: units on a scale] — The maximum score is 30 points. Score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.
  units on a scale | 28.6 (1.2) | 27.5 (2.5) | 28.2 (2.1)
Intrinsic Motivation Inventory, score out of 7 [Mean (Standard Deviation); unit: units on a scale] — The mean of the 7 items is the summary score for the Intrinsic Motivation - Interest and Enjoyment Subscale (Min possible 1, Max possible 7). Higher number indicates higher interest/enjoyment.
  units on a scale | 5.6 (1.0) | 5.6 (1.1) | 5.6 (1.1)
Chakrabarty Grade, score out of 100 [Mean (Standard Deviation); unit: units on a scale] — The sum of all items is the score (Min possible -104, Max possible 100). Higher score indicates more favorable residual limb health.
  units on a scale | 77.3 (16.2) | 82.4 (15.0) | 79.8 (15.6)
Comorbidity Index, score out of 20 [Mean (Standard Deviation); unit: units on a scale] — The comorbidity index is a sum of 18 comorbidities (Min possible 0, Max possible 18). Higher score indicates higher comorbidity.
  units on a scale | 6.1 (2.7) | 7.1 (2.3) | 6.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Timed Up-and-Go Test
Description: Performance-based physical function test able to predict falls for people with lower limb amputation. The TUG test time is taken from rising from a chair, walking 3 meters, turning, walking back and sitting down. Continuous scale; higher time indicates lower physical function, higher likelihood of falls.
Time Frame: Baseline, 12-weeks, and 24 weeks
Population: 38 (35 men, 3 women; 19 INT, 19 CTL) enrolled. 1 INT and 1 CTL lost to follow-up. 36 participants assessed at all time points. Two CTL at 12 weeks and 2 CTL,1 INT at 24 weeks completed questionnaires only.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
seconds
  Baseline | 19.4 [14.8 to 23.9] | 20.7 [15.6 to 25.7]
  12-Week: number analyzed (Participants) | 18 | 16
  12-Week | 18.2 [13.4 to 22.9] | 18.8 [13.6 to 24.1]
  24-week: number analyzed (Participants) | 17 | 16
  24-week | 16.7 [12.1 to 21.3] | 21.3 [16.0 to 26.7]
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.87, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.38, Mixed Models Analysis

2. Secondary Outcome: Two-Minute Walk Test
Description: Performance-based physical function test measures total number of meters walked in two minutes on a level walkway.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
meters
  Baseline | 86.9 [76.9 to 96.9] | 84.4 [73.2 to 95.6]
  12-Week: number analyzed (Participants) | 18 | 16
  12-Week | 88.5 [77.6 to 99.3] | 83.3 [71.3 to 95.3]
  24-Week: number analyzed (Participants) | 17 | 16
  24-Week | 99.8 [89.6 to 110.0] | 84.0 [72.0 to 96.1]
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.75, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.11, Mixed Models Analysis

3. Secondary Outcome: Five Meter Walk Test
Description: Performance-based physical function test measures the time to walk 5 meters at the participant's "normal, everyday pace".
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: meters/second
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
meters/second
  Baseline | 0.78 [0.69 to 0.88] | 0.76 [0.66 to 0.87]
  12-Week: number analyzed (Participants) | 18 | 16
  12-Week | 0.96 [0.86 to 1.06] | 0.83 [0.71 to 0.94]
  24-Week: number analyzed (Participants) | 17 | 16
  24-Week | 0.97 [0.87 to 1.06] | 0.86 [0.75 to 0.98]
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.11, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.23, Mixed Models Analysis

4. Secondary Outcome: Prosthesis Evaluation Questionnaire - Mobility Section
Description: Self-report physical function questionnaire measures capacity to perform a list of specific functional tasks (e.g., walking upstairs, getting in and out of a vehicle. Scores range from being unable or hardly able (0) to having no problems (4). An average score across the 12-item questionnaire was used in the analysis. Lower numbers indicate less difficulty.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 2.2 [1.7 to 2.8] | 2.1 [1.5 to 2.8]
  12-Week | 2.6 [2.0 to 3.2] | 2.0 [1.3 to 2.6]
  24-Week | 2.7 [2.1 to 3.3] | 2.4 [1.7 to 3.0]
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.27, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.58, Mixed Models Analysis

5. Secondary Outcome: Houghton Scale
Description: Self-report physical function questionnaire. The outcome is the sum of scores from each item (min 0, max 12). A higher score indicates higher self-report of physical function with the prosthesis.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 0.64 (0.15) | 0.62 (0.23)
  12-Week | 0.69 (0.28) | 0.69 (0.24)
  24-Week | 0.77 (0.18) | 0.65 (0.27)
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.83, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.13, Mixed Models Analysis

6. Secondary Outcome: Patient-Specific Function Scale
Description: Self-report physical function questionnaire. The outcome is the average score for up to five participant-identified activities on a scale from 0-10 (min 0, max 10). Higher score indicates greater ability to perform functional activities.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 3.3 (1.8) | 3.5 (1.9)
  12 weeks | 5.7 (2.6) | 5.1 (2.3)
  24 weeks | 6.9 (2.3) | 5.3 (2.3)
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.02, t-test, 2 sided

7. Secondary Outcome: Physical Activity Step Counts
Description: Instrumented physical activity measure, average step counts per day
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: average steps per day
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
average steps per day
  Baseline | 1305 [726 to 1883] | 1369 [724 to 2014]
  12-Week: number analyzed (Participants) | 18 | 16
  12-Week | 2439 [1844 to 3035] | 1512 [849 to 2175]
  24-Week: number analyzed (Participants) | 17 | 16
  24-Week | 2294 [1716 to 2873] | 1510 [840 to 2180]
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.03, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.06, Mixed Models Analysis

8. Secondary Outcome: Self-Efficacy in Managing Chronic Disease Questionnaire
Description: Scale range is 1-10. The score for the scale is the mean of the six items, using a ten point scale. Higher number indicates higher self-efficacy.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 7.6 [7.1 to 8.3] | 7.5 [6.8 to 8.2]
  12-Week | 7.8 [7.2 to 8.4] | 7.9 [7.2 to 8.6]
  24-Week | 8.1 [7.5 to 8.7] | 7.5 [6.8 to 8.2]
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.62, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.40, Mixed Models Analysis

9. Secondary Outcome: World Health Organization Disability Assessment Scale
Description: Scores ranging from 1 (no difficulty) to 5 (extreme difficulty/cannot do). Overall disability was calculated by summing the scores for the 12 items; higher scores indicated greater disability (score range: 12-60).
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 26.2 [22.9 to 29.6] | 27.5 [23.7 to 31.3]
  12-Week | 24.2 [20.9 to 27.6] | 25.3 [21.5 to 29.2]
  24-Week | 21.6 [18.2 to 25.0] | 25.3 [21.4 to 29.1]
Statistical Analysis 1: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 12-week test; Test type: Superiority; p = 0.96, Mixed Models Analysis
Statistical Analysis 2: Comparison: Exercise, Activity, and Self-management vs Home and Phone Visit; Test null hypothesis that there is no difference between groups from baseline to 24-week test; Test type: Superiority; p = 0.35, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Exercise, Activity, and Self-management | Home and Phone Visit
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 4/19 | 9/19
Other Adverse Events (participants affected / at risk) | 14/19 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise, Activity, and Self-management (N=19) | Home and Phone Visit (N=19)
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) — Pneumonia
Hospitalization (Infections and infestations) | 1 (1) | 5 (7)
Hospitalization (Endocrine disorders) | 1 (2) | 1 (1) — Hypoglycemia
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Hallucinations
Hospitalization (General disorders) | 0 (0) | 1 (1) — Opiod Overdose
Hospitalization (General disorders) | 0 (0) | 1 (1) — Edema
Hospitalization (General disorders) | 0 (0) | 1 (1) — Increased medical management
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise, Activity, and Self-management (N=19) | Home and Phone Visit (N=19)
Fall (General disorders) | 10 (16) | 8 (12)
Wound Infection (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Foot Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size limited statistical power to identify group differences in secondary outcomes. CTL group exercise behavior only tracked step count. No direct measurement of intervention fidelity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-01-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT01929018/Prot_000.pdf
  • Statistical Analysis Plan (2014-01-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT01929018/SAP_001.pdf